CLINICAL TRIAL: NCT00977366
Title: Pilot Study Investigating Central Sensitisation of the Cough Reflex in Subjects With Chronic Cough and Healthy Volunteers
Brief Title: Neurophysiology of Cough Reflex Hypersensitivity
Acronym: NOTCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Collaborators: JP Moulton Charitable Foundation (Other); Medical Research Council (Other Government)
Responsible Party: Principal Investigator, Jacky Smith, MRC Clinician Scientist/Honorary Respiratory Consultant, University of Manchester
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 09/H1004/21
Record Dates: First submitted 2009-09-14; First posted 2009-09-15 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Cough; Healthy Controls
MeSH Terms: conditions — Cough | interventions — Hydrochloric Acid; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hydrochloric acid infusion (Active Comparator)
  Interventions: Other: Hydrochloric acid (0.15 molar)
- Saline (Placebo Comparator)
  Interventions: Other: Saline

INTERVENTIONS:
Other: Hydrochloric acid (0.15 molar) — Hydrochloric acid (0.15 molar) will be infused in to the lower oesophagus through a distal infusion port located at the tip of an oesophageal stimulation catheter.
  Arms: Hydrochloric acid infusion
Other: Saline — Normal saline will be infused in to the lower oesophagus through a distal infusion port located at the tip of an oesophageal stimulation catheter.
  Arms: Saline

SUMMARY:
Central sensitisation is an increase in the excitability of nerves within the central nervous system, which can lead to heightened sensitivity to certain stimuli. This process is involved in some chronic pain conditions e.g. migraines and non-cardiac chest pain. Recent work by our group suggests central sensitisation may be an important mechanism leading to chronic cough.

The main questions in this study include:

1. Can the investigators induce temporary central sensitisation of the cough reflex in healthy volunteers for testing of new medications?
2. Can the investigators demonstrate exaggerated sensitisation in patients with chronic cough (indicating these patients are already centrally sensitised)?

In animal studies, acid infusion into the gullet (oesophagus) is able to induce central sensitisation of the cough reflex. Acid infusion into the oesophagus has also been shown to induce central sensitisation in human healthy volunteers, increasing the sensitivity to pain on the front of the chest but this study did not test the the cough reflex. Using human participants, the investigators plan to test whether acid infusion into the oesophagus increases the sensitivity of the cough reflex in healthy volunteers and also patients complaining of chronic cough.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers inclusion:

* Over 18 years
* Measurable cough reflex sensitivity - required as is the primary end-point
* No current or past history of chronic cough or chronic respiratory disease

Chronic Cough Patients inclusion:

* Over 18 years
* Chronic persistent cough (> 8 weeks) despite investigation and/or treatment trials for cough variant asthma/post-nasal drip and gastro-oesophageal reflux
* Normal chest radiograph - primary respiratory cause for cough excluded
* Normal lung function - primary respiratory cause for cough excluded Measurable cough reflex sensitivity - required as primary end-point

Exclusion Criteria:

* Recent upper respiratory tract infection (<4 weeks) - this can lead to increased sensitivity of the cough reflex which resolves as the infection settles
* Pregnancy/breast-feeding - unknown effects of oesophageal acid infusion
* Current smokers or ex-smokers with < 6 month abstinence or history > 20 pack years - smoking can alter the sensitivity of the cough reflex
* Opiate or ACE inhibitor use or centrally acting medication - can alter the cough reflex sensitivity
* Symptomatic gastro-oesophageal reflux, post-nasal drip or asthma (chronic cough cohort may have been treated for these in the past but cough did not resolve) - these conditions are known to cause cough and alter cough reflex sensitivity
* Significant ongoing chronic respiratory/cardiovascular/gastro-intestinal/haematological/ neurological/psychiatric illness. We are aiming to recruit healthy volunteers and chronic cough patients who are otherwise healthy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2010-03; Primary Completion 2012-09 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Effect of oesophageal acid infusion on cough reflex sensitivity in chronic cough patients compared to healthy controls. | baseline, immediatley after infusion, 90 minutes post infusion, 180 minutes post infusion, 24 hours after baseline
  Outcome measures include; cough reflex sensitivity, pain threshold measures, 24 hour objective cough rate

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Woodcock, Prof, Principal Investigator — The University of Manchester
Locations (1):
- University Hospital of South Manchester, Manchester, United Kingdom